CLINICAL TRIAL: NCT04139174
Title: Assessment of Root Parallelism Following Orthodontic Treatment in Adolescent vs Adult Patients Treated With Maxillary First Premolar Extraction: Observational -Analytical Study
Brief Title: Assessment of Root Parallelism Following Orthodontic Treatment in Adolescent vs Adult Patients Treated With Maxillary First Premolar Extraction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina adly kaldas, principal investigator, Cairo University
Other Study IDs: orthodontics 3-3-4
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Frequency of Root Paralellism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adolescent group: Panoramic radiographs of finished orthodontic cases will be collected after fulfilling the inclusion and exclusion criteria. Then the collected data will be divided into two groups according to age either adolescent (12-18 years old) or adult group (after 18 years old).
  measurements will be done on the radiograph using digital software.
  Interventions: Procedure: first premolar extraction and complete canine retraction.
- adult group: Panoramic radiographs of finished orthodontic cases will be collected after fulfilling the inclusion and exclusion criteria. Then the collected data will be divided into two groups according to age either adolescent (12-18 years old) or adult group (after 18 years old).
  measurements will be done on the radiograph using digital software.
  Interventions: Procedure: first premolar extraction and complete canine retraction.

INTERVENTIONS:
Procedure: first premolar extraction and complete canine retraction. — measurements on panoramic radiograph will be done after first premolar extraction and complete canine retraction.

SUMMARY:
Panoramic radiographs of finished orthodontic cases will be collected after fulfilling the inclusion and exclusion criteria. Then the collected data will be divided into two groups according to age either adolescent (12-18 years old) or adult group (after 18 years old).

in the panoramic views the long axes of canines and second premolar will be traced digitally using Digital softwares (microDicom vierwer Simeo Antonov Stoykov 0.7.7) & (IC Measure 2.0.0.161).

The objective of this study is to assess the root parallelism between maxillary canines and second premolars in adolescents versus adults group of patients requiring maxillary first premolar extraction during the orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults group of Patients (above 18 years old). .
* Adolescent group of patients (from 12 to 18 years old).
* Extraction of permanent maxillary first premolar in at least one quadrant.
* Same head position at scanning time.
* Same machine: Orthopantomograph Planmeca Promax 2P (Planmeca USA) with a kilovoltage of 55 to 85 and an exposure time of 15 seconds at a focal distance of 46 cm.
* Same type of bracket (Roth prescription, slot size #22).
* Full set of teeth (not necessarily including third molars)

Exclusion Criteria:

* Systematic diseases.
* non extraction cases.
* severe divergence or convergence between roots of maxillary canine and second premolar.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the collected data will be divided into two groups according to age either adolescent (12-18 years old) or adult group (after 18 years old).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of Good Root Parallelism | 8 months
  root paralellism between canine and second premolar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oshagh M, Momenidanaei S, Sardarian A, Alipour A, Roeinpeykar M, Khaksar Y. Root Parallelism of Canine and Second Premolar. 2014;3(3):176-81.
- [Result] Mayoral G. Treatment results with light wires studied by panoramic radiography. Am J Orthod. 1982 Jun;81(6):489-97. doi: 10.1016/0002-9416(82)90428-6. PMID 6960734